CLINICAL TRIAL: NCT04693377
Title: Cryoablation Combined With Stereotactic Body Radiation Therapy for the Treatment of Painful Bone Metastases
Brief Title: Cryoablation Combined With Stereotactic Body Radiation Therapy for the Treatment of Painful Bone Metastases, the CROME Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-1234; NCI-2020-07368 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1234 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-13; First posted 2021-01-05 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Prostate Carcinoma; Metastatic Renal Cell Carcinoma; Metastatic Sarcoma; Metastatic Thyroid Gland Carcinoma; Metastatic Urothelial Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Melanoma; Prostatic Neoplasms; Carcinoma, Renal Cell; Sarcoma; Thyroid Neoplasms; Carcinoma, Transitional Cell | interventions — Cryosurgery; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (SBRT) (Active Comparator): Patients undergo stereotactic body radiation therapy for 1 fraction.
  Interventions: Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy
- Arm B (cryoablation, SBRT) (Experimental): Patients undergo cryoablation. Within 10 days after cryoablation, patients undergo stereotactic body radiation therapy for 1 fraction. Alternatively, patients may receive stereotactic body radiation therapy initially, followed by cryoablation."
  Interventions: Procedure: Cryosurgery; Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Cryosurgery — Undergo cryoablation
  Other Names: Ablation, Cryo; Cryoablation; cryosurgical ablation
  Arms: Arm B (cryoablation, SBRT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Stereotactic Body Radiation Therapy — Undergo stereotactic body radiation therapy
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This trial compares cryoablation combined with stereotactic body radiation therapy to stereotactic body radiation therapy alone to see how well they work in treating patients with pain from cancer that has spread to the bones (bone metastases). Bone is a common site of metastasis in advanced cancer, and bone metastases often result in debilitating cancer-related pain. The current standard of care to treat painful bone metastases is radiation therapy alone. However, many patients do not get adequate pain relief from radiation therapy alone. Another type of therapy that may be used to provide pain relief from bone metastases is cryoablation. Cryoablation is a procedure in which special needles are inserted into the tumor site. These needles grow ice balls at their tips to freeze and kill cancer cells. The goal of this trial is to compare how well cryoablation in combination with radiation therapy works to radiation therapy alone when given to cancer patients to provide pain relief from bone metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of cryoablation in combination with stereotactic body radiation therapy (SBRT) or SBRT only for the treatment of painful bone metastases.

SECONDARY OBJECTIVES:

I. To assess for narcotics utilization by daily morphine equivalent dose. II. To assess duration of pain response reported by International Pain Response Criteria.

III. To assess for local tumor control. IV. To assess for changes in patient quality of life with Brief Pain Inventory (BPI) score.

V. To assess for adverse event rates. VI. To assess incidence and severity of adverse events/toxicity. VII. To assess technical success for cryoablation.

EXPLORATORY OBJECTIVE:

I. To investigate the local microenvironmental changes following SBRT and cryoablation combined with SBRT to bone metastases.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo stereotactic body radiation therapy for 1 fraction.

ARM B: Patients undergo cryoablation. Within 10 days after cryoablation, patients undergo stereotactic body radiation therapy for 1 fraction.

After completion of study treatment, patients are followed up at 1, 2, 3, 4, 8, 12, 16, 20, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a primary diagnosis of malignancy and radiographic evidence of bone metastases. Eligible tumor histologies include the following malignancies with low alpha/beta ratios: renal cell carcinoma, urothelial carcinomas, castration-resistant prostate cancer, sarcoma, thyroid carcinoma, colorectal carcinoma, and melanoma
* A target lesion the meets the following criteria:

  * The target lesion must be amenable to both cryoablation and SBRT, as determined by the study principal investigators (PIs)
  * The target lesion must be =< 7cm
  * The pain due to the target lesion must be at least 4/10 based on the BPI pain scale
  * Pain from the metastatic site must correlate with an identifiable tumor on computed tomography (CT), magnetic resonance imaging (MRI), or ultrasound (US) imaging
* Life expectancy >= 3 months
* Platelet count > 50,000/mm^3 within 6 weeks of screening
* International normalized ratio (INR) < 1.5 within 6 weeks of screening
* If taking antiplatelet or anticoagulation medication, it must be able to be discontinued 48 hours prior to the procedure or at the discretion of the PI (e.g., aspirin, ibuprofen, low molecular weight heparin [LMWH] preparations)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%) within 6 weeks of screening
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization. Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization
* All lines of prior systemic therapy are permissible. Standard concurrent chemotherapy, immunotherapy, or targeted therapy are permissible
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior locoregional therapy to target lesion, including ablation of any modality, embolization, radiation, or surgery
* Patient may not be receiving any other investigational agents. Standard concurrent chemotherapy, immunotherapy, or targeted therapy will be allowed
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing women; women of childbearing potential unless using effective contraception as determined by the investigator
* Target lesions that involve the spinal column or calvarium
* Absolute neutrophil count < 1000 mm^3 within 6 weeks of screening
* Active infection
* Presence of confirmed pathologic fracture at the target lesion not amenable to percutaneous stabilization
* Lesions that involve a weight-bearing long bone of the lower extremity with the tumor causing > 50% loss of cortical bone. Lesions involving the hands and feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain response | At 12 weeks post-treatment
  Defined as complete or partial response as reported by the International Pain Response Criteria at the site of the treated bone metastasis based on the BPI pain score and daily morphine equivalent (MEDD). Will be summarized separately for each treatment arm with associated 95% exact confidence intervals.

SECONDARY OUTCOMES:
Daily morphine equivalent (MEDD) | Baseline, assessed up to 24 weeks post-treatment
Duration of response | Up to 24 weeks post-treatment
  Will be assessed by performing area under the curve (AUC) analysis of Brief Pain Inventory (BPI) pain scores.
Local control | Up to 24 weeks post-treatment
  Will be determined by imaging evidence of residual viable tumor. Standard of care cross-sectional imaging and bone scintigraphy will be performed at 3 month intervals.
Rate and severity of adverse and serious related adverse events | Within 30 days of the last study treatment
  Point estimates and two-sided 95% confidence intervals will be generated for procedural related adverse events.
Technical success for cryoablation | Up to 24 weeks post-treatment
  Will be determined by identifying on intra-procedural imaging when the leading edge of the ice successfully extends beyond the tumor margin by at least 5 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul A Sheth, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org